CLINICAL TRIAL: NCT03134534
Title: The Study of Robotic-assisted Thoracoscopic Lobectomy Versus Video-assisted Thoracoscopic Lobectomy for Non-small Cell Lung Cancer (RVlob)
Brief Title: Robot-assisted vs VATS Lobectomy for NSCLC
Acronym: RVlob
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Hecheng Li M.D., Ph.D, Professor, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTS-002
Record Dates: First submitted 2017-04-15; First posted 2017-05-01 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Pulmonary Neoplasm
Keywords: lobectomy; robot-assisted thoracoscopic surgery; lung cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VATS group (Other): Surgical procedure: VATS lobectomy
  Interventions: Procedure: VATS lobectomy
- RATS group (Other): Surgical procedure: RATS lobectomy
  Interventions: Procedure: RATS lobectomy

INTERVENTIONS:
Procedure: VATS lobectomy — a minimal invasive surgical types for NSCLC: VATS lobectomy
  Arms: VATS group
Procedure: RATS lobectomy — a minimal invasive surgical types for NSCLC: RATS lobectomy
  Arms: RATS group

SUMMARY:
Robot-assisted thoracoscopic surgery (RATS) was widely used in thoracic surgery, the surgical safety and feasibility of RATS lobectomy for NSCLC has been confirmed. However, the oncological long-term outcomes of RATS lobectomy has not been studied by randomized controlled trial, the purpose of this study is to determine whether RATS lobectomy would be as effective as VATS lobectomy on short-term and long-term outcomes.

DETAILED DESCRIPTION:
Video-assisted thoracoscopic surgery (VATS) lobectomy is recommended for non small cell lung cancer (NSCLC) with surgical indications in China, its oncological long-term outcomes has been widely approved. As a new form of VATS, robot-assisted thoracoscopic surgery (RATS) was widely used in thoracic surgery, the 3D vision and flexible robot arm were helpful for surgeons to perform precise operations, and RATS was reported to bring extra benefits to patients. The surgical safety and feasibility of RATS lobectomy for NSCLC has been confirmed. However, the oncological long-term outcomes of RATS lobectomy has not been studied by randomized controlled trial. so we designed this randomized controlled trial to determine whether RATS lobectomy would be as effective as VATS lobectomy on short-term and long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. surgical indication for lobectomy;
2. minimal invasive surgery;
3. ASA (American Society of Anesthesiologists) stage: I-III;
4. sign the informed consent. -

Exclusion Criteria:

1. benign tumor or nodule;
2. present of other malignancy;
3. preoperative chemotherapy, radiotherapy, targeted therapy. -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
3-year overall survival (OS) | 3 year after surgery
  OS at 3 year after surgery
Lymph node counts | postoperative in-hospital stay up to 30 days
  overall lymph node counts, number of stations dissected, and number of lymph nodes in each lymph node station

SECONDARY OUTCOMES:
3-year disease-free survival (DFS) | 3 year after surgery
  DFS at 3 year after surgery
1-year overall survival (OS) | 1 year after surgery
  OS at 1 year after surgery
1-year disease-free survival (DFS) | 1 year after surgery
  DFS at 1 year after surgery
R0 rate | postoperative in-hospital stay up to 30 days
  R0 radical rate
margin state | postoperative in-hospital stay up to 30 days
  positive margin rate
operative time | postoperative in-hospital stay up to 30 days
  the time of operation
blood loss | postoperative in-hospital stay up to 30 days
  blood loss in the operation
conversion rate | postoperative in-hospital stay up to 30 days
  the rate of conversion to open surgery in the operation
operative accident event | postoperative in-hospital stay up to 30 days
  the accident event happened in operative
30-day mortality | postoperative in-hospital stay up to 30 days
  30-day mortality after surgery
length of stay (LOS) | postoperative in-hospital stay up to 30 days
  length of stay in hospitalization
postoperative complications | postoperative in-hospital stay up to 30 days
  mainly include: pneumonia, arrhythmia, incision infection, vocal cord paralysis, trachea cannula
quality of life (QOL) at 3 month | at 3 month after surgery
  QOL, WHOQOL-BREF

OTHER OUTCOMES:
total hospitalization expenditures | postoperative in-hospital stay up to 30 days
  cost in hospital

CONTACTS AND LOCATIONS:
Overall Officials: He-Cheng Li, doctor, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai JiaoTong University School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Li C, Chen X, Wang X, Guo W, Zhang Y, Chen F, Li H. Single-Port Robotic-Assisted Approach in Thoracic Surgery: A Prospective Real-World Study. Interdiscip Cardiovasc Thorac Surg. 2025 Jul 3;40(7):ivaf161. doi: 10.1093/icvts/ivaf161. PMID 40658465
- [Derived] Niu Z, Cao Y, Du M, Sun S, Yan Y, Zheng Y, Han Y, Zhang X, Zhang Z, Yuan Y, Li J, Zhang Y, Li C, Han D, Du H, Guo W, Chen K, Xiang J, Zhu L, Che J, Hang J, Ren J, Lerut T, Abbas AE, Lin J, Jin R, Li H. Robotic-assisted versus video-assisted lobectomy for resectable non-small-cell lung cancer: the RVlob randomized controlled trial. EClinicalMedicine. 2024 Jul 12;74:102707. doi: 10.1016/j.eclinm.2024.102707. eCollection 2024 Aug. PMID 39105193
- [Derived] Jin R, Zhang Z, Zheng Y, Niu Z, Sun S, Cao Y, Zhang Y, Abbas AE, Lerut T, Lin J, Li H. Health-Related Quality of Life Following Robotic-Assisted or Video-Assisted Lobectomy in Patients With Non-Small Cell Lung Cancer: Results From the RVlob Randomized Clinical Trial. Chest. 2023 Jun;163(6):1576-1588. doi: 10.1016/j.chest.2022.12.037. Epub 2023 Jan 5. PMID 36621757
- [Derived] Jin R, Zheng Y, Yuan Y, Han D, Cao Y, Zhang Y, Li C, Xiang J, Zhang Z, Niu Z, Lerut T, Lin J, Abbas AE, Pardolesi A, Suda T, Amore D, Schraag S, Aigner C, Li J, Che J, Hang J, Ren J, Zhu L, Li H. Robotic-assisted Versus Video-assisted Thoracoscopic Lobectomy: Short-term Results of a Randomized Clinical Trial (RVlob Trial). Ann Surg. 2022 Feb 1;275(2):295-302. doi: 10.1097/SLA.0000000000004922. PMID 33938492